CLINICAL TRIAL: NCT00228592
Title: A Phase II, Multicenter, Randomized, Open-Label, Dose-Ranging, Parallel Group Study to Compare the Anti-Viral Effects, Pharmacokinetics and Safety of HepeX-Bä, a Mixture of Two Monoclonal Antibodies, as Compared to Hepatitis B Immune Globulin in Patients Who Have Received Hepatic Allografts for Treatment of End-Stage Liver Disease Due to Hepatitis B Virus Infection
Brief Title: HepeX-B in Post Hepatic Allografts for Treatment of End Stage Liver Disease Due to Hepatitis B Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HepeX-B 2003-12
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2007-02

CONDITIONS: Hepatitis B; Liver Transplantation
MeSH Terms: conditions — Hepatitis B | interventions — hepatitis B hyperimmune globulin

INTERVENTIONS:
Drug: HepeX-B
Drug: Hepatitis B Immune Globulin (HBIg)

SUMMARY:
The purpose of this study is to compare the use of HepeX-B versus HBIg, two anti-viral drugs, in patients who have received liver transplants due to liver failure caused by Hepatitis B infection. Patients will be evaluated over a 6 month to 1.5 year period to evaluate whether or not the drugs prevent the Hepatitis B virus from infecting the new liver.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients who are 18 years of age or older,
* Patients who are at least 6 months post first orthotopic liver transplantation (living or cadaveric donor) for treatment of end-stage liver disease due to HBV infection,
* Patients who have received HBIg since transplantation and are on a stable regimen (i.e., same dose and frequency) for at least the 3 months immediately preceding study entry (Day 1),
* Patients who have received treatment with an inhibitor of HBV polymerase for at least the 3 months immediately preceding study entry (Day 1),
* Patients with undetectable HBsAg and HBV DNA concentrations on two consecutive tests at least 1 week apart during the screening period,
* Female patients who are of childbearing potential, and males whose partners are women of childbearing potential, are required to use adequate contraception, and
* Patients who are able to provide written informed consent.
* Patients who successfully complete the initial 20-week treatment in the core trial are eligible for the 52-week extension phase.

Exclusion Criteria:

* Women who are pregnant or breastfeeding,
* Patients who have received another organ transplant that requires immunosuppression,
* Patients who are co-infected with hepatitis delta virus (HDV), hepatitis C virus (HCV) and/or human immunodeficiency virus (HIV),
* Patients with clinical conditions or diseases, which, in the judgment of the investigator, would place the patient at undue risk, interfere with study participation, or confound the results of the study, and/or
* Patients who have participated in clinical studies in the 3 months prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Rustgi, MD, Principal Investigator — Metropolitan Liver Diseases/ Gastroenterology Center
Locations (20):
- United States (12):
  - UCLA, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - UCSF, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska, Omaha, Nebraska
  - Mt. Sinai, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Metropolitan Liver Diseases/Gastroenterology Center, Fairfax, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
- Centre Hepato-Biliaire Hospital Paul Brousse, Paris, France
- Humbolt University Virchow Clinic Dept. Viceral and Transplant Surgery, Berlin, Germany
- Israel (3):
  - Hadassah University Hospital, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Auckland City Hospital, Auckland, New Zealand
- Hospital La Fe Servicio de Medicina Degestiva, Valencia, Spain
- Royal Free Hospital, London, United Kingdom